CLINICAL TRIAL: NCT00503503
Title: Safety and Efficacy From Large Scale All Cases Surveillance for Etanercept in Japan
Brief Title: Study Evaluating the Efficacy of Enbrel (Etanercept) in Subjects in Japan
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0881Y1-4460
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Enbrel (etanercept)

SUMMARY:
The objective of this surveillance is to determine the following items in all patients receiving Enbrel for a certain period after marketing: 1) unlabeled adverse events, 2) onset (frequency, severity and other details) of adverse events, 3) factors considered to affect the safety, and 4) the efficacy of Enbrel. Moreover, the onset (frequency, severity and other details) of the followings will be key issues of this surveillance:Infection (tuberculosis, opportunistic infection, etc.), autoimmune diseases, cardiac failure, malignant tumor, interstitial pneumonia, demyelinating disorders, pancytopenia, aplastic anemia and application site reactions.

ELIGIBILITY:
Inclusion Criteria

· Patients with rheumatoid arthritis [only those refractory to the previous treatment]

Ages: 11 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Koike T, Harigai M, Inokuma S, Inoue K, Ishiguro N, Ryu J, Takeuchi T, Tanaka Y, Yamanaka H, Fujii K, Freundlich B, Suzukawa M. Postmarketing surveillance of the safety and effectiveness of etanercept in Japan. J Rheumatol. 2009 May;36(5):898-906. doi: 10.3899/jrheum.080791. Epub 2009 Mar 30. PMID 19332630